CLINICAL TRIAL: NCT00006031
Title: Randomized Prospective Trial Comparing Radioactive Seed Localized Breast Biopsy to Needle Localized Breast Biopsy
Brief Title: Comparison of Two Types of Biopsy in Patients With Breast Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MCC-12114; NCI-G00-1808 (Other: NCI)
Record Dates: First submitted 2000-07-05; First posted 2004-04-02 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Breast Cancer
Keywords: biopsy; radioactive seed; nonpalpable lesions
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I: Radioactive Seed Localized Breast Biopsy (Active Comparator): Arm I: Patients undergo radiographic placement of a radioactive seed (either iodine I 125 or palladium Pd 103) into the suspicious lesion. Patients then undergo surgery to remove the lesion along with the seed and a small margin of surrounding breast tissue followed 3 months later by a postoperative mammogram.
  Interventions: Procedure: Low dose radioactive seed followed by surgery and mammogram
- Arm II: Needle Localized Breast Biopsy (Active Comparator): Arm II: Patients undergo a needle localized breast biopsy with a specimen x-ray.
  Interventions: Procedure: Needle localized breast biopsy with specimen x-ray

INTERVENTIONS:
Procedure: Needle localized breast biopsy with specimen x-ray
  Arms: Arm II: Needle Localized Breast Biopsy
Procedure: Low dose radioactive seed followed by surgery and mammogram — either iodine I 125 or palladium Pd 103
  Arms: I: Radioactive Seed Localized Breast Biopsy

SUMMARY:
RATIONALE: Biopsy is the removal of cells or tissue for examination under a microscope. It is not yet known which type of breast biopsy is more effective for diagnosing breast lesions.

PURPOSE: Randomized diagnostic trial to compare the effectiveness of two different types of biopsy in patients who have breast lesions that cannot be felt upon examination.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the effect of low dose radioactive seed localized breast biopsy versus needle localized breast biopsy on operative time and tissue loss in patients with nonpalpable breast lesions. II. Compare the cost effectiveness of these diagnostic methods in these patients. III. Demonstrate that radioactive seed localization allows for elimination of specimen x-ray in these patients. IV. Demonstrate that radioactive seeds may be placed safely for 1-7 days prior to surgical removal in these patients.

OUTLINE: This is a randomized study. Patients are randomized to one of two diagnostic arms. Arm I: Patients undergo radiographic placement of a radioactive seed (either iodine I 125 or palladium Pd 103) into the suspicious lesion. Patients then undergo surgery to remove the lesion along with the seed and a small margin of surrounding breast tissue followed 3 months later by a postoperative mammogram. Arm II: Patients undergo a needle localized breast biopsy with a specimen x-ray.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Suspicious nonpalpable breast lesion requiring breast biopsy for diagnosis OR Nonpalpable breast lesion that is not amenable to core needle biopsy or advanced breast biopsy instrumentation (ABBI) excision Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Menopausal status: Not specified Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Not pregnant

PRIOR CONCURRENT THERAPY: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 1999-11; Primary Completion 2001-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Tissue Loss Rates for Each Arm | 18 months
  Compare the effect of low dose radioactive seed localized breast biopsy versus needle localized breast biopsy on tissue loss in patients with nonpalpable breast lesions.
Operative Time Rates in Each Group | 18 months
  Compare the effect of low dose radioactive seed localized breast biopsy versus needle localized breast biopsy on operative time in patients with nonpalpable breast lesions.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events for Each Group | 18 months
  Review of adverse events utilizing Common Toxicity Criteria (CTC) V3.

CONTACTS AND LOCATIONS:
Overall Officials: Charles E. Cox, MD, FACS, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States